CLINICAL TRIAL: NCT05558956
Title: Total Body PET-CT Imaging of Prostate Cancer Using Illuccix (Kit for the Preparation of Ga-68 PSMA-11 Injection)
Brief Title: Total Body PET-CT Imaging of Prostate Cancer Using Illuccix
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BAMF Health (Other)
Collaborators: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BAMF-2022-03
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose (Experimental): 3 mCi dose of 68Ga-PSMA-11 (Illuccix) and a total body PET-CT scan for 4-6 min scan time.
  Interventions: Drug: illuccix 68Ga-PSMA-11 Total Body PET-CT
- High dose (Experimental): 7 mCi dose of 68Ga-PSMA-11 (Illuccix) and a total body PET-CT scan for 4-6 min scan time.
  Interventions: Drug: illuccix 68Ga-PSMA-11 Total Body PET-CT

INTERVENTIONS:
Drug: illuccix 68Ga-PSMA-11 Total Body PET-CT — Illuccix (kit for the preparation of gallium Ga 68 gozetotide injection) 68Ga-PSMA-11

SUMMARY:
Illuccix will be used per the prescribing instructions for PET-CT imaging on the United Imaging scanner uEXPLORER to establish a standard scanning protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male ≥ 18 years of age
3. Patients meeting clinical need for Illuccix PET scan:

   1. Patients with suspected metastasis who are candidates for initial definitive therapy
   2. Patients with suspected recurrence based on elevated serum prostate-specific antigen (PSA) level
4. Patient is physically able to lay flat for the PET-CT procedure

Exclusion Criteria:

1. Assessment by the Investigator as unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the imaging quality using low dose and high dose Ga-68 PSMA-11 at various scan lengths. | 3 months
  In modulating the dose and scan time, including reconstitution of the images, we will identify optimal protocol for use of Illuccix on total body PET/CT through evaluation of image quality at variable dose and scan length.

CONTACTS AND LOCATIONS:
Locations (1):
- BAMF Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No